CLINICAL TRIAL: NCT05188404
Title: Cannabis Use Among Older Adults: Potential Risks and Benefits to an Aging Population
Brief Title: Aging and Marijuana: Benefits, Effects, and Risks
Acronym: AMBER
Status: Completed | Type: Observational
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Other Study IDs: 1R01AG066698 (NIH)
Record Dates: First submitted 2021-12-10; First posted 2022-01-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Cannabis Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cannabis Users: Older adults (60 and up) who report pain, sleep problems, and/or negative mood (anxiety and/or depression) and who desire to use cannabis for these issues (n=300)
  Interventions: Behavioral: Choice of cannabis product
- Cannabis Non-users: Older adults (60 and up) who report pain, sleep problems, and/or negative mood (anxiety and/or depression) and do NOT desire to use cannabis for these issues (n=50)

INTERVENTIONS:
Behavioral: Choice of cannabis product — Participants choose and purchase their own cannabis product
  Groups: Cannabis Users

SUMMARY:
Investigators will gather data on both the beneficial and harmful effects of edible cannabis of varying composition (THC-only vs. CBD-only vs. THC+CBD), and will examine the process by which older adult cannabis users decide what type of cannabis product is preferred.

DETAILED DESCRIPTION:
Older adults are currently the fastest growing group of cannabis users in the U.S, and are more likely to use cannabis for medicinal purposes (e.g., pain, trouble sleeping, depression/anxiety) than for recreational purposes, despite having little data to guide their decisions about what type of product to use. This project utilizes a patient-centered observational design to recruit and assess older adults who are interested in using cannabis compared to a control group who is not interested in cannabis use. Investigators will gather data on both the beneficial and harmful effects of edible cannabis of varying composition (THC-only vs. CBD-only vs. THC+CBD), and will examine the process by which older adult cannabis users decide what type of cannabis product is preferred.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years of age
* Able to provide informed consent
* Cannabis Users: Must not currently use cannabis more than 7 times per month and not for pain, sleep, depression or anxiety in the past 6 months
* Cannabis Non-users: Should NOT have used cannabis in the past year and have not used regularly (e.g., more than weekly) for more than one year in the past 20 years
* Cannabis Users: Must be interested in using cannabis for at least one of the following complains: pain, sleep problems, depression, anxiety
* Non-users: Must NOT be interested in using cannabis but have at least one of the following complaints: pain, sleep problems, depression, anxiety
* Cannabis users: must be comfortable using edible cannabis and having a mobile laboratory (Dodge van) parked at their home
* Female participants must be postmenopausal
* Comfortable reading and writing in English
* Planning to stay in the Boulder/Denver area for the next month
* Must be comfortable with blood draws

Exclusion Criteria:

* Blood alcohol level > 0 at screening (to sign consent form)
* Report of other drug use (cocaine, opiates, methamphetamine) in the past 90 days or fail urine screen for any of these drugs
* Past or current diagnosis of psychosis
* Current use of antipsychotic medications
* Heavy drinking; Alcohol Use Disorder Identification Test (AUDIT) test score >8
* Inability/discomfort/unwillingness with getting in and out of the mobile laboratory van
* History of vertigo or falls within the past six months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults experiencing problems with pain, sleep, depression or anxiety who either wish to use cannabis or who do not wish to cannabis
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Patient Global Impression of Change | 1-month, 2 months, 3 months, 4 months
  Self report of whether symptoms have improved, gotten worse, or stayed the same
Change in FACT-Cog | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether cognitive function has improved, gotten worse, or stayed the same
Change in Rey Auditory Verbal Learning Task | Baseline, 1-month
  Test of whether working memory has improved, gotten worse, or stayed the same
Balance Task | 1-month
  Stability with eyes closed and eyes open
Change in Activities Specific Balance Confidence Scale | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether confidence in balance has improved, gotten worse, or stayed the same

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scale | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether depression, anxiety and stress have improved, gotten worse, or stayed the same
Change in PROMIS Sleep Disturbance | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether sleep quality has improved, gotten worse, or stayed the same
Change in PROMIS Fatigue | Baseline, 1-month, 2 months, 3 months, 4 months
  Measure of whether experience of fatigue has improved, gotten worse, or stayed the same
Change in PROMIS Pain Interference | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether the extent to which pain interferes with daily life activities has improved, gotten worse, or stayed the same
Change in pain Intensity past 7 days | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether intensity of pain has improved, gotten worse, or stayed the same
Current Pain Intensity | 1-month
  Self-reported intensity of pain right now
Addiction Research Center Inventory Marijuana Survey | 1-month
  Acute subjective effects of cannabis
Drug Effects Questionnaire | 1-month
  Acute subjective effects of cannabis
Profile of Mood States | 1-month
  Acute mood effects of cannabis
Change in PROMIS Global Health | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether general health and functioning has improved, gotten worse, or stayed the same
Change in Polypharmacy | Baseline, 1-month, 2 months, 3 months, 4 months
  Measure of whether number and dosage of current medications has improved, gotten worse, or stayed the same
Change in Online Timeline Follow-back Assessment | Baseline, 1-month, 2 months, 3 months, 4 months
  30-day retrospective report of substance use (cannabis, alcohol, other drugs); measure of whether substance use has improved, gotten worse, or stayed the same
Change in Marijuana Consumption Questionnaire | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether frequency and quantity of cannabis use changes over time or stays the same

OTHER OUTCOMES:
Change in Blood Cannabinoids and Endocannabinoids | Baseline, 1-month
  Quantitation of major and minor cannabinoids and endocannabinoids in blood; measure of whether cannabinoid levels change over time
Change in Neurofilament Light | Baseline, 1-month
  Quantitation of neuronal damage in blood; measure of whether damage change over time
Change in Expectancies about Cannabis | Baseline, 1-month, 2 months, 3 months, 4 months
  Self-report of whether opinions about the health effects of cannabis has improved, gotten worse, or stayed the same
Change in Flanker Inhibitory Control and Attention task | Baseline, 1-month
  Measure of whether inhibition has improved, gotten worse, or stayed the same

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No